CLINICAL TRIAL: NCT06702020
Title: VIS Opti-K Vision Improvement for Presbyopes
Acronym: VIS Opti-K 002
Status: Active, not recruiting | Type: Observational
Sponsor: VIS, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VIS Opti-K-Presbyopia #002
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Presbyopia Correction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The VIS Opti-K device and procedure were used to provide vision improvement to patients with presbyopia.

DETAILED DESCRIPTION:
The VIS Opti-K device was used to irradiate the cornea with light that changed corneal shape.

ELIGIBILITY:
Inclusion Criteria:

Female or male Any race 40 years of age or older Presbyopia

Exclusion Criteria:

None

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had documented presbyopia and a need for near vision improvement
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2007-03-13 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Uncorrected distance and near visual acuities | Up to 24 months post-treatment
  Uncorrected distance and near visual acuities are measured using ETDRS or similar charts.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Berry, PhD, Principal Investigator — VIS, Inc.

IPD SHARING:
Plan to Share IPD: No
Privacy

REFERENCES:
- See also: VIS, Inc website — http://www.viscorrect.com